CLINICAL TRIAL: NCT04085978
Title: A Retrospective Analysis of the Effects of a Hypoglycemia Protocol With Glucose Gel on NICU Admission
Brief Title: Effects of a Hypoglycemia Protocol With Glucose Gel on Neonatal Intensive Care Unit (NICU) Admission
Status: Terminated | Type: Observational
Why Stopped: The standard of care had changed during our wait for the Program Letter of Agreement between Phoenix Children's Hospital and Banner to administering IV glucose in the newborn nursery so we weren't able to meet our objective.
Sponsor: Pediatrix (Other)
Collaborators: Banner University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 501938027
Record Dates: First submitted 2019-09-05; First posted 2019-09-11 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Hypoglycemia; Neonatal Hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre implementation of hypoglycemia protocol with glucose gel: All neonates born at Banner University Hospital during January 01, 2014 - November 30, 2016 who qualify for hypoglycemia protocol
- Post implementation of hypoglycemia protocol with glucose gel: All neonates born at Banner University Hospital during January 01, 2018 - November 30 2018 who qualify for hypoglycemia protocol

SUMMARY:
Evaluate if the implementation of a hypoglycemia protocol with glucose gel has reduced the NICU admission rate of neonates with low-acuity neonatal hypoglycemia.

DETAILED DESCRIPTION:
This project will evaluate various aspects of infants with hypoglycemia admitted to the Neonatal Intensive Care Unit (NICU) pre- and post- implementation of a hospital-wide hypoglycemia protocol with oral glucose gel. Subjects will be matched by gestational age (GA), birth weight rounded to the nearest half kilogram, ethnicity, gender, maternal age, maternal diabetes status, maternal parity, maternal ethnicity, and mode of delivery. Retrospective data will be reviewed including neonatal and maternal demographics and NICU medical course data. The results of this study can inform intended and unintended consequences of the instituted protocol.

ELIGIBILITY:
Inclusion Criteria:

* All neonates born at Banner University Hospital during January 01, 2014 - November 30, 2016 and January 01, 2018 - November 30 2018 who qualify for hypoglycemia protocol.

Exclusion Criteria:

* Neonates <34 weeks gestational age or with birth weight less than 2000 grams.
* Infants with serious congenital malformation
* Infants with a terminal disorder.

Min Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To detect a 130% increase in NICU length of stay with power of 0.8, the investigators calculated a sample size of 400 subjects with 200 subjects before and after implementation. It is estimated that the data collection period is roughly over the course of one year, with the assumption that not all neonates with hypoglycemia will meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Mean NICU length of stay rounded to the day | 30 days
  Mean NICU length of stay rounded to the day
Mean maximum glucose infusion rate | 30 days
  Mean maximum glucose infusion rate

SECONDARY OUTCOMES:
Assess for complications | 30 days
  - Number of neonates identified to have any type of infection
Assess for weight loss | 30 days
  - Maximum weight loss as percent below birth weight during NICU admission
Evaluate for persistent symptomatic or asymptomatic hypoglycemia | 30 days
  * Number of neonates with symptomatic hypoglycemia
  * Number of neonates with asymptomatic hypoglycemia
Number of neonates who received formula | 30 days
  Time to gain back to birthweight (if occurred while in-house), rounded to day of life
Number of neonates with any breastfeeding during hospitalization | 30 days
  Time to gain back to birthweight (if occurred while in-house), rounded to day of life
Number of neonates with breastfeeding at time of discharge | 30 days
  Time to gain back to birthweight (if occurred while in-house), rounded to day of life

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Martin, MD, Principal Investigator — Pediatrix
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States